CLINICAL TRIAL: NCT03655613
Title: A Phase 1/2 Dose Escalation and Expansion Study of Combination APL-501 or Nivolumab With APL-101 in Locally Advanced or Metastatic Hepatocellular and Renal Cell Carcinoma
Brief Title: APL-501 or Nivolumab in Combination With APL-101 in Locally Advanced or Metastatic HCC and RCC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to administrative reasons.
Sponsor: Apollomics (Australia) Pty. Ltd. (Industry)
Collaborators: Apollomics Inc. (formerly CBT Pharmaceuticals, Inc.) (Unknown); Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APOLLO
Record Dates: First submitted 2018-07-17; First posted 2018-08-31 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Hepatocellular Carcinoma; Renal Cell Carcinoma
Keywords: Immunotherapy; PD-1 inhibitor; c-Met inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: (Phase 1) 3+3 dose escalation (Phase 2) Simon two-stage Minimax design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Hepatocellular Carcinoma (Experimental): PD-1 inhibitor (APL-501) 3 mg/kg intravenously every 2 weeks + c-Met inhibitor (APL-101) 150 mg or 200 mg administered twice daily continuously until documented disease progression, discontinuation due to toxicity withdrawal of consent or the study ends
  Interventions: Biological: APL-501; Drug: APL-101
- Arm B: Renal Cell Carcinoma (Experimental): PD-1 inhibitor (nivolumab) 3 mg/kg or 240 mg intravenously every 2 weeks + c-Met inhibitor (APL-101) 300 mg or 400 mg administered twice daily continuously until documented disease progression, discontinuation due to toxicity withdrawal of consent or the study ends
  Interventions: Drug: APL-101; Biological: Nivolumab

INTERVENTIONS:
Biological: APL-501 — Humanized IgG4 monoclonal antibody against programmed death receptor-1 (PD-1)
  Other Names: genolimzumab; GB226; CBT-501
  Arms: Arm A: Hepatocellular Carcinoma
Drug: APL-101 — Oral specific c-Met inhibitor
  Other Names: bozitinib; vebreltinib; CBT-501
Biological: Nivolumab — Fully human IgG4 monoclonal antibody against PD-1
  Other Names: Opdivo
  Arms: Arm B: Renal Cell Carcinoma

SUMMARY:
Study Design and Investigational Plan:

This is an open-label Phase 1/2 study to assess the safety and tolerability of combination PD-1 inhibitor (APL-501 or nivolumab) administered concomitantly with c-Met inhibitor (APL-101), to determine the recommended Phase 2 dose of the combination, and to obtain preliminary efficacy in HCC or RCC subjects with advanced or metastatic disease that have not been previously treated with a PD 1 inhibitor or a c-Met inhibitor. HCC subjects will receive the combination APL-501 plus APL-101 while RCC subjects will receive the combination nivolumab plus APL-101. In Phase 1, mandatory archival or fresh tumor biopsies will be collected. In Phase 2, a mandatory fresh tumor biopsy will be required for study entry and another fresh biopsy will be collected between Cycles 2 and 4. The frequency of administration of PD-1 inhibitors will be every 2 weeks starting in Cycle 1 on Day 8 and Day 22 of a 35-day cycle with all subsequent cycles on Day 1 and Day 15 of 28-day cycles. APL-101 will be administered orally every 12 hours continuously on an empty stomach.

DETAILED DESCRIPTION:
For each potential subject, there is a 28-day screening and eligibility assessment period before enrollment; the first dose of study treatment will be administered on Day 1 of Cycle 1 (C1D1) (Safety population). Subjects will continue to receive their assigned treatment throughout the study until the occurrence of confirmed disease progression [progressive disease (PD)] by irRECIST, death, unacceptable treatment-related toxicity, or until the study is closed by the Sponsor. During the treatment period, study visits will occur on Day 1, Day 2, Day 8, Day 15, Day 22 of Cycle 1 and Day 1 and Day 15 of every subsequent cycle. Subjects who experience a response [Complete Response (CR), Partial Response (PR)] ≥ 2 cycles, PD 1 plus APL-101 combination will be continued until disease progression based on irRECIST. Subjects should receive a minimal of 2 cycles of PD-1 and APL-101 for adequate evaluation of response (Evaluable population). Discontinuation of PD-1 and APL-101 should occur upon determination of disease progression as determined by irRECIST, intolerable toxicity or when the risk/benefit ratio is no longer beneficial for the subjects as determined by the Principal Investigator, or upon subject withdrawal of consent. Upon permanent discontinuation of study treatment, there is a Treatment Termination visit and three monthly follow-up visits for a 90-day safety follow-up visit period. Subjects who drop out before they complete the first cycle of combination treatment for reasons other than toxicity will be replaced

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent.
2. Men and women 18 years of age or older.
3. Histologically confirmed advanced or metastatic hepatocellular carcinoma that progressed while receiving at least one previous line of systemic therapy, including sorafenib, or who are intolerant of or refused sorafenib treatment following progression on standard therapy including surgical and/or local regional therapies, or standard therapy considered ineffective, intolerable, or inappropriate or for which no effective standard therapy is available.
4. Histologically confirmed advanced or metastatic renal cell carcinoma with clear cell component who received one or two prior lines of antiangiogenic therapy in addition to no more than three previous regimens of systemic therapy including cytokines and cytotoxic chemotherapy agents.
5. Disease according to irRECIST that can be reliably and consistently followed.
6. Documented disease progression during or after the last treatment regimen and within 6 months before study enrollment.
7. Tumor amenable to tumor biopsy and subject agreeable to tumor biopsy at study entry and during therapy with study treatment.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
9. Acceptable organ function.

Exclusion Criteria:

1. History of severe hypersensitivity to mAbs, excipients of the APL-501, nivolumab, or APL-101.
2. History of receiving treatment with any c-Met signaling pathway inhibitor (marketed or investigational agents).
3. Prior therapy with anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibody (or any other antibody targeting T cell co-stimulation pathways).
4. Unwilling to swallow orally administered medication whole.
5. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption (e.g., Crohn's, ulcerative colitis, active inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).
6. Documented and/or known history of human immunodeficiency virus (HIV) for HCC and RCC subjects, or historical seropositive results consistent with active infection for hepatitis C virus (HCV) or hepatitis B virus (HBV) (RCC only).
7. HCC subjects receiving active antiviral therapy for HCV.
8. Active co-infection with HBV and HCV.
9. Active co-infection with HBV and hepatitis D virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (Phase 1) | Cycle 1 (up to 35 days)
  Dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Adverse events | First dose up to 90 days post last dose (up to approximately 2 years)
  Toxicity grading will be performed in accordance with NCI CTCAE, version 4.0. including immune related adverse events (irAEs)
Drug discontinuation due to adverse events | First dose up to 90 days post last dose (up to approximately 2 years)
  Toxicity grading will be performed in accordance with NCI CTCAE, version 4.0. including immune related adverse events (irAEs)
Overall Response Rate | Duration of study, performed at baseline, then every 8 weeks until objective disease progression (up to approximately 2 years)
  Tumor response will be assessed by immune related Response Evaluation Criteria in Solid Tumors (irRECIST)
Time to Response | Duration of study, first dose to first response (up to approximately 2 years)
  Time to response is the time from first dose to date of first response (Partial response or Complete response)
Progression Free Survival | Duration of study, performed at baseline, then every 8 weeks until objective disease progression at 6, 12, 18 and 24 months (up to approximately 2 years)
  Progression free survival will be collected on all enrolled subjects, defined as the time from first dose to death from any cause or first observed disease progression
Overall Survival | Duration of study, performed every 8 weeks from enrollment to death from any cause at 6, 12, 18, 24 months (up to approximately 2 years)
  Overall survival will be estimated using the Kaplan-Meier method with the follow-up starting at the initiation of therapy until date of death

CONTACTS AND LOCATIONS:
Overall Officials: Scott Houston, Study Director — Apollomics (Australia) Pty. Ltd.
Locations (9):
- Australia (8):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Crown Princess Mary Cancer Centre, Westmead, New South Whales
  - Ashford Cancer Center, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Sunshine Hospital, Saint Albans, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Afffinity Clinical Research, Perth, Western Australia
- Auckland City Hospital, Auckland, New Zealand

REFERENCES:
- See also: Company website for Apollomics Inc. — http://www.apollomicsinc.com/